CLINICAL TRIAL: NCT06157736
Title: Microbiome in the Acute Stage of New Onset Paediatric Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: APC Microbiome Ireland (Unknown)
Responsible Party: Principal Investigator, Professor Colin Hawkes, Associate Professor of Pediatrics, University College Cork
Other Study IDs: Acute T1D
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Urine Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children with newly diagnosed T1D
- Controls: Healthy siblings of cases

SUMMARY:
The goal of this observational study is to learn more about the microbiome and metabolome of children with type 1 diabetes (T1D). The main questions it aims to answer are:

1. Do the microbiome and metabolome play a role in the onset and presentation of T1D?
2. How do the microbiome and metabolome evolve during the early stages of T1D?
3. Are there are differences in the microbiome or metabolome of children who present with diabetic ketoacidosis (DKA) versus those who present without DKA, and between those who present with mild, moderate or severe DKA?
4. Is there an association between the microbiome or metabolome and glycaemic control during the first year of diagnosis?
5. Is there an association between the microbiome or metabolome and beta cell reserve after one year of T1D disease?

DETAILED DESCRIPTION:
T1D is caused by autoimmune-mediated destruction of pancreatic beta cells. This leads to a complete deficiency of insulin. Individuals diagnosed with T1D require life-long exogenous insulin replacement to achieve glucose homeostasis and, ultimately, to survive. Although there is an underlying genetic predisposition to developing T1D, the trigger is multifactorial and likely includes environmental factors.

Several large cohort studies have identified differences in the microbiome in those with T1D compared to healthy controls and suggested that it may have a role in the pathogenesis of T1D. It is not yet clear if changes in the microbiome are involved in the pathogenesis of beta-cell destruction or are an effect of the disease state.

When children present with T1D for the first time, their blood glucose levels are elevated. Some children will present with life threatening DKA in which there is metabolic dysfunction and, in some cases, end organ damage.

This study will examine the microbiome and metabolome of children with newly diagnosed T1D during their initial hospital admission, and describe the changes that occur in the microbiome and metabolome as these individuals are commenced on insulin and return to normal glucose homeostasis.

The study will also compare the microbiome and metabolome of children presenting with and without DKA to establish if there are particular patterns of microbial diversity which are more common in one group. The study also aims to establish if there is an association between the microbiome or metabolome and glycaemic control during the first year of T1D diagnosis. The study will also investigate associations between the microbiome and metabolome, and beta cell reserve after the first year of T1D disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with newly diagnosed T1D.
2. Aged between 6 months and 18 years at their first study visit.
3. Consent provided by parent/guardian to participate in this study.
4. Age dependent assent or consent obtained for participants aged 6-18 years

Exclusion Criteria:

1. Individuals who have a known diagnosis of inflammatory bowel disease or another medical condition which the study team deems might interfere with the microbiome.
2. Individuals with complex medical or behavioural needs that would deem the participant unable to participate in the study.
3. Have a significant acute or chronic co-existing illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic) or any condition which contraindicates entry to the study according to the investigator's judgement.
4. Participants who are receiving treatment involving experimental medications.
5. If the participant took part in a recent experimental trial, the trial must have been completed not less than 30 days prior to participation in this study.
6. Have a malignant disease or any concomitant end-stage organ disease

Ages: 6 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children aged between 6 months and 18 years who are admitted to hospital with a new diagnosis of T1D will be assessed for eligibility for enrolment to this study.
  Healthy siblings will be assessed for eligibility to be enrolled as controls in this study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Describe evolution of the microbiome and metabolome during the early stages of new onset T1D | 52 weeks
  Microbiome biodiversity in cases vs controls

CONTACTS AND LOCATIONS:
Overall Officials: Colin Hawkes, Principal Investigator — University College Cork
Locations (1):
- Cork University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kennedy EC, Ross FC, O'Shea CA, Lavelle A, Ross P, Dempsey E, Stanton C, Hawkes CP. Observational study protocol: the faecal microbiome in the acute stage of new-onset paediatric type 1 diabetes in an Irish cohort. BMJ Open. 2025 Jan 30;15(1):e089206. doi: 10.1136/bmjopen-2024-089206. PMID 39890137